CLINICAL TRIAL: NCT00960102
Title: Children's Bilateral Cochlear Implantation in Finland: a Prospective, Controlled, Multicenter Study
Brief Title: Children's Bilateral Cochlear Implantation in Finland
Acronym: FinBiCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); Hospital District of Helsinki and Uusimaa (Other); University of Helsinki (Other); Oulu University Hospital (Other); University of Oulu (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Heikki Lopponen, M.D.,Prof., Kuopio University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5551819
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Deafness; Hearing Loss
Keywords: cochlear implantation; hearing aid
MeSH Terms: conditions — Deafness; Hearing Loss | interventions — Cochlear Implants; Hearing Aids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- bilateral cochlear implant (Active Comparator)
  Interventions: Device: cochlear implant
- cochlear implant and hearing aid (Active Comparator)
  Interventions: Device: cochlear implant; Device: hearing aid
- bilateral hearing aid (Active Comparator)
  Interventions: Device: hearing aid

INTERVENTIONS:
Device: cochlear implant — Multichannel Nucleus cochlear implant
  Arms: bilateral cochlear implant; cochlear implant and hearing aid
Device: hearing aid — Phonak hearing aid
  Arms: bilateral hearing aid; cochlear implant and hearing aid

SUMMARY:
The purpose of this study is to evaluate short and long term outcomes (benefits and side-effects) of bilateral cochlear implantation and bilateral hearing aid rehabilitation in Finnish children.

ELIGIBILITY:
Inclusion Criteria:

* Congenital severe or profound bilateral hearing impairment
* No functional benefit from conventional hearing aids (minimum 3 months trial)
* Radiologically (CT,MRI) patent inner ears and normal central auditory pathways
* Family is motivated for rehabilitation programme and gives a written consent
* Finnish or Swedish as the primary language in the home

Exclusion Criteria:

* A child has an additional anomaly or disability that may affect to his/her functional or neurological development
* Inner ear anomaly
* Mother's pregnancy duration less than 32 weeks

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of auditory performance skills of bilaterally or bimodally implanted children or children with bilateral hearing aids | Various time points up to 5 years hearing age

SECONDARY OUTCOMES:
To compare post-operative speech perception ability, language acquisition, and speech production | Various time points up to 5 years hearing age
To compare speech recognition performance | Various time points up to 5 years hearing age
Quality of life and functional communicative performance assessed by parental proxy measures, and health economical assessment | Various time points up to 5 years hearing age
To evaluate operative and post-operative complications, side-effects and device failures | Various time points up to 5 years hearing age
To evaluate the differences in balance function | at 3 and 5 year age

CONTACTS AND LOCATIONS:
Overall Officials: Heikki J Löppönen, M.D.,Prof., Study Director — Department of Otorhinolaryngology, Institute of Clinical Medicine, Kuopio University and Kuopio University Hospital, Finland; Taina T Välimaa, Ph.D., Principal Investigator — Faculty of Humanities, Logopedics, University of Oulu, Finland
Locations (5):
- Finland (5):
  - Department of Otorhinolaryngology, Helsinki University Hospital, Helsinki
  - Department of Otorhinolaryngology, Kuopio University Hospital, Kuopio
  - Department of Otorhinolaryngology, Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Department of Otorhinolaryngology, Turku University Hospital, Turku

REFERENCES:
- [Derived] Valimaa TT, Kunnari S, Aarnisalo AA, Dietz A, Hyvarinen A, Laitakari J, Mykkanen S, Rimmanen S, Salonen J, Sivonen V, Tennila T, Tsupari T, Vikman S, Virokannas N, Laukkanen-Nevala P, Tolonen AK, Tuohimaa K, Lopponen H. Spoken Language Skills in Children With Bilateral Hearing Aids or Bilateral Cochlear Implants at the Age of Three Years. Ear Hear. 2022 Jan/Feb;43(1):220-233. doi: 10.1097/AUD.0000000000001092. PMID 34260435